CLINICAL TRIAL: NCT03006653
Title: Understanding Daily Fluctuations in Self-Regulation
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Collaborators: Cornell University (Other); Sage Bionetworks (Other)
Responsible Party: Sponsor
Other Study IDs: 16-693
Record Dates: First submitted 2016-12-27; First posted 2016-12-30 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Impulsive Behavior; Self-Regulation
MeSH Terms: conditions — Impulsive Behavior; Self-Control

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Assessment only — Mobile ecological assessment only.

SUMMARY:
Understanding Daily Fluctuations in Self-Regulation, also known as the Digital Marshmallow Test (DMT), is a collaboration by Northwell Health, Cornell Tech, and Sage Bionetworks. Funded by the Robert Wood Johnson Foundation, this is a pioneering study to advance the science in identifying and helping individuals who act on short-term temptations, despite long-term consequences. Using Apple's ResearchKit(™) and Android's ResearchStack applications, the Digital Marshmallow Test will leverage the powerful capabilities of the smartphone to examine impulsivity using a range of game-like tasks and sensor capabilities within the mobile phone. Across studies, more impulsive individuals are significantly more likely to suffer from obesity, Type II Diabetes, substance abuse, gambling problems, suicidal behaviors, and increased criminality among many other problems. Early self-report studies reveal a relationship between the inability to delay gratification and different patterns of mobile phone use. This will be the first study to develop non-invasive mobile methods to identify and help those at greatest risk for impulsive responding before serious problems occur.

DETAILED DESCRIPTION:
Poor self-regulation and impulsivity are underlying symptoms of numerous mental health problems such as obesity, substance abuse, Attention Deficit Hyperactivity Disorder (ADHD), gambling, binge eating, bipolar disorder, borderline personality disorder, and suicidal behaviors. This makes it one of the most important personal and public health intervention targets. The classic Marshmallow Test done by Mischel and colleagues determined that the inability to delay gratification in childhood was predictive of lower Scholastic Aptitude Test (SAT) scores and higher BMI in adulthood. However, assessments of impulsivity and poor self-regulation are rarely included in routine medical care because of time and financial constraints.

The mobile phone has changed our ability to assess and intervene with individuals remotely, providing an avenue for ambulatory diagnostic testing and just-in-time adaptive interventions that can be accessed by billions of people. Newer methods of assessment using the mobile phone, including Apple's ResearchKit, provide the opportunity for powerful assessments of impulsivity beyond simple self-report. To date, there have been no measures of impulsivity integrated into ResearchKit or any mobile application, aside from the beta version that the investigators recently built, nor has the research community explored the possibilities of passive impulsivity assessment using mobile analytics embedded in all phones. There is preliminary evidence that mobile analytics, such as latency to respond to a text, can predict personality traits associated with impulsivity such as extroversion and neuroticism, and self-report studies reveal that there is a direct relationship between the inability to delay gratification and different patterns of mobile phone use. These studies highlight potential power of mobile phenotyping as a ubiquitous measure of health determinants in billions of people by using passive data that doesn't require user participation. However, foundational research is needed to validate assessments, build adaptive tools, and include individual differences self-regulation capacity as well as interventions to improve regulation in the discussion.

The investigators propose to test a new diagnostic self-regulation mobile assessment tool app. The application built in Apple's ResearchKit(™) and Android's ResearchStack(™) includes a self-report assessment, three continuous performance tasks, and passive data collection developed for in-person use.

The goal is that by differentiating between high and low impulsive people using mobile assessment tools, the investigators identify those at greatest risk for self-regulation problems. Individuals higher in impulsivity have less self-control when faced with short-term temptations regardless of their knowledge of the consequences of these choices. This would be the first step in developing a completely remote measurement tool for this purpose.

The primary goal of this exploratory project is to develop and validate a mobile application to test impulsivity remotely, and test how self-report indicators of impulsivity via mobile assessment correlate with objective impulsivity tests on the mobile phone.

Because this is an exploratory study, the investigators are looking at how often participants use the mobile app in the real-world and how the tasks perform over time once they leave the laboratory. In addition, the investigators will test the validity of the measures over time.

ELIGIBILITY:
Inclusion Criteria:

* be fluent and able to read in English at the eighth grade level (self-report and consent form quiz),
* be between the ages of 18 and 75 (self-report, age in demographics),
* be willing to provide informed consent, and
* own a mobile smartphone (iOS or Android) and are willing to receive and respond to text messages.

Exclusion Criteria:

* are pregnant or breast feeding,
* present with significant substance use which is defined as greater than once weekly use in the past month (for any substance other than alcohol, nicotine or caffeine) or greater than 21 standard alcoholic drinks per week for women and 24 for men,
* present with a serious psychiatric illness or suicide risk as measured by previous inpatient treatment, medications for psychosis or recent suicidality; a current self-reported or clinician determined diagnosis of Major Depression or past or present bipolar disorder, delusional disorder or schizophrenia, and/or
* are unable to understand research study procedures as evidenced a score of less than 4 out of 5 on the consent form quiz.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participant must be fluent and able to read in English at the eight grade level, be between the ages of 18 and 75, be willing to provide informed consent, and own a mobile smartphone (iOS or Android) and are willing to receive and respond to text messages.
Sampling Method: Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Impulsivity | 21 Days
  Daily assessment of impulsivity.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Muench, PhD, Principal Investigator — Northwell Health
Locations (1):
- Center for Addiction Services and Personalized Interventions Research (CASPIR), Great Neck, New York, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared. No plan in place.

REFERENCES:
- [Background] Billieux J, van der Linden M, Rochat L. The role of impulsivity in actual and problematic use of the mobile phone. Applied Cognitive Psychology 22: 1195-1210, 2008.
- [Background] Lazer D, Pentland A, Adamic L, Aral S, Barabasi AL, Brewer D, Christakis N, Contractor N, Fowler J, Gutmann M, Jebara T, King G, Macy M, Roy D, Van Alstyne M. Social science. Computational social science. Science. 2009 Feb 6;323(5915):721-3. doi: 10.1126/science.1167742. No abstract available. PMID 19197046
- [Derived] Wen H, Sobolev M, Vitale R, Kizer J, Pollak JP, Muench F, Estrin D. mPulse Mobile Sensing Model for Passive Detection of Impulsive Behavior: Exploratory Prediction Study. JMIR Ment Health. 2021 Jan 27;8(1):e25019. doi: 10.2196/25019. PMID 33502330
- [Derived] Sobolev M, Vitale R, Wen H, Kizer J, Leeman R, Pollak JP, Baumel A, Vadhan NP, Estrin D, Muench F. The Digital Marshmallow Test (DMT) Diagnostic and Monitoring Mobile Health App for Impulsive Behavior: Development and Validation Study. JMIR Mhealth Uhealth. 2021 Jan 22;9(1):e25018. doi: 10.2196/25018. PMID 33480854